CLINICAL TRIAL: NCT06202690
Title: Single-POrt Robotic Versus Video-assisted Thoracic Surgery Anatomical Pulmonary Resection for Patients With Non-small Cell Lung Cancer (SPORTS Study): a Single-center, Single-blinded, Randomized Controlled Trial
Brief Title: SP Robotic Versus VATS Anatomical Pulmonary Resection for Patients With NSCLC
Acronym: SPORTS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Korea University Guro Hospital (Other)
Responsible Party: Principal Investigator, Hyun Koo Kim, Professor, Korea University Guro Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2023GR0429
Record Dates: First submitted 2023-11-09; First posted 2024-01-11 (Actual); Last update posted 2024-01-11 (Actual); Status verified 2024-01

CONDITIONS: Robotics; Lung Cancer
Keywords: sing-port surgery, robotic-assisted thoracic surgery, lung cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Intervention Model Description: This trial is a single-center, single blinded, randomized controlled trial). Participants will be randomized in a 1:1 ratio to either to single-port video-assisted thoracoscopic surgery (SP-VATS) or single-port robotic-assisted thoracic surgery (SP-RATS).
Who Masked: Participant
Masking Description: The principal investigator will explain the study at the time of consent for the surgery. Written consent will be obtained by the principal investigator or a sub-investigator. Once eligibility for surgery is confirmed, randomization will take place within 4 weeks prior to the surgery. Participants will be randomized in a 1:1 ratio to either SP-RATS or SP-VATS using a website software randomization system. While the surgeon will be informed of the group allocations, participants will remain unaware (maintaining a single-blind approach) until the completion of the follow-up period
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SP-RATS (Active Comparator): SP-RATS Arm: 145 patients, single-port anatomical pulmonary resection will be performed using the SP robotic system. A 4-cm single incision will be made below the subcostal margin. A chest tube will be inserted in same incision.
  Interventions: Procedure: Single-port robotic-assisted thoracic surgery
- SP-VATS (Placebo Comparator): SP-VATS Arm: 145 patients, single-port anatomical pulmonary resection was performed using VATS. A 4-cm incision will be made at 5th intercostal space on the anterior or posterior axillary line. A chest tube will be inserted in same incision.
  Interventions: Procedure: Single-port video-assisted thoracoscopic surgery

INTERVENTIONS:
Procedure: Single-port robotic-assisted thoracic surgery — All patients : 145 patients Single-port anatomical pulmonary resection(segmentectomy, lobectomy) with a complete mediastinal lymph node dissection will be performed using the SP robotic system.
  A 4-cm single incision will be made below the subcostal margin. A chest tube will be inserted in same incision.
  Other Names: SP-RATS
  Arms: SP-RATS
Procedure: Single-port video-assisted thoracoscopic surgery — All patients : 145 patients Single-port anatomical pulmonary resection(segmentectomy, lobectomy) with a complete mediastinal lymph node dissection will be performed using the VATS.
  A 4-cm single incision will be made at 5th intercostal space. A chest tube will be inserted in same incision.
  Other Names: SP-VATS
  Arms: SP-VATS

SUMMARY:
Single-POrt Robotic-assisted thoracic surgery versus single-port video-assisted Thoracic Surgery major pulmonary resection for patients with non-small cell lung cancer (SPORTS trial): a single-center, a single blinded, randomized controlled trial

DETAILED DESCRIPTION:
Investigators initially began single-port robotic thoracic surgery using the SP robotic system for simple procedures, such as thymectomy and mediastinal mass excision. As their expertise grew, they expanded to more complex procedures, including major pulmonary resection and esophagectomy. However, the long-term outcomes of SP robotic anatomical pulmonary resection using the SP robotic system have not yet been studied.

The aim of this study is to compare the short-term and long-term outcomes of SP robotic anatomical pulmonary resection using the SP robotic system with those of single-port video-assisted thoracoscopic surgery (SP-VATS) anatomical pulmonary resection.

This trial is a single-center, single-blinded, randomized controlled trial. Participants will be randomized at a 1:1 ratio to either single-port video-assisted thoracoscopic surgery (SP-VATS) or single-port robotic thoracic surgery.

ELIGIBILITY:
Inclusion Criteria:

* Candidate for anatomical pulmonary resection (segmentectomy or lobectomy) via minimally invasive thoracic surgery (RATS or VATS) for patient with non-small cell lung cancer or suspected malignant lesion.
* Age ≥ 18 years
* Patients who can comply with the requirements of the clinical trial and who, or their legal representatives, provide written consent before the start of the clinical trial
* Patients with the nationality of South Korea
* American Society of Anesthesiologists score 1-3.
* Clinical stage I, II or IIIa non-small cell lung cancer (NSCLC)

Exclusion Criteria:

* Patients who require surgery for accompanying other organ diseases
* Tumor invasion into the chest wall, diaphragm, another lobe or diaphragm
* Patients who are considered unsuitable based on the researcher's judgment
* Patients with cognitive impairments who are unable to understand the instructions and informed consent of this study
* Patients who specifically desire a certain surgical method (robotic, thoracoscopic, open thoracotomy)
* Patients who previously undergone a thoracic surgical procedure in the hemithorax to be operated on
* Pathological results other than NSCLC (ex, benign nodules, metastatic lung cancer, SCLC)
* Patients who received neoadjuvant therapy.
* Candidate for pneumonectomy, bilobectomy, lobectomy plus segmentectomy, non-anatomic resection (ex, wedge resection).
* History of other cancers in the past 5 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 290 (Estimated)
Dates: Start 2024-01-09 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2031-06-30 (Estimated)

PRIMARY OUTCOMES:
Postoperative complications | Postoperative complications : within 30 days after surgery
  complications will be classified according to Clavien-Dindo classfication
Questionnaires for HRQOL of life (EQ-5D-5L) at month 3 | at month 3 after surgery
  Questionnaires for HRQOL of life (EQ-5D-5L) will be administered at months 3.
Questionnaires for HRQOL of life (EQ-VAS) at month 3 | at month 3 after surgery
  Questionnaires for HRQOL of life (EQ-5D-5L, EQ-VAS) will be administered at months 3.
Postoperative pain | during hospitalization
  Pain levels were assessed and recorded using the VAS score more than three times daily during the hospitalization period.

SECONDARY OUTCOMES:
Questionnaires for HRQOL of life (EQ-5D-5L) | At 2 weeks before surgery, and at 1 month, 6 months, and 12 months, as well as at years 2, 3, 4, and 5 after surgery.
  Questionnaires for HRQOL of life (EQ-5D-5L, EQ-VAS) will be administered at 2 weeks before surgery, and at 1 month, 6 months, and 12 months, as well as at years 2, 3, 4, and 5 after surgery.
Questionnaires for HRQOL of life (EQ-VAS) | At 2 weeks before surgery, and at 1 month, 6 months, and 12 months, as well as at years 2, 3, 4, and 5 after surgery.
  Questionnaires for HRQOL of life (EQ-5D-5L, EQ-VAS) will be administered at 2 weeks before surgery, and at 1 month, 6 months, and 12 months, as well as at years 2, 3, 4, and 5 after surgery.
Questionnaires for HRQOL of life (LCQ) | at 1 month, 3 months, and 6 months after surgery.
  Questionnaires for HRQOL of life (LCQ) will be administered at 1 month, 3 months, and 6 months after surgery.
Perioperative outcomes (Conversion rate) | during hospitalization
  Conversion rate = conversion to open thoracotomy / total number of surgery
Perioperative outcomes (number of lymph nodes harvested) | during hospitalization
  Total number of lymph nodes harvested during the surgical procedure.
Perioperative outcomes (total operative time) | during hospitalization
  the time taken from skin incision to completion of skin closure
Perioperative outcomes (duration of chest tube drainage, postoperative hospital stays) | during hospitalization
  duration of chest tube drainage: the time from the date of the operation to the date of chest tube removal
  postoperative hospital stays: the time from the date of the operation to the date of discharge
Perioperative outcomes (transfusion rate) | within 30 days after surgery.
  The transfusion rate was defined as the percentage of patients who received an allogeneic blood transfusion within 30 days after surgery.
Perioperative outcomes (estimated blood loss ) | during surgery
  estimated measurement of intraoperative blood loss (ml)
5-year overall survival and disease-free survival | 5 years
  Overall survival (OS) is defined as the time from randomization to death. Disease-free survival (DFS) is defined as the time from randomization to recurrence of tumor or death.

IPD SHARING:
Plan to Share IPD: No